CLINICAL TRIAL: NCT03889613
Title: Pillcam Crohn's Capsule for Monitoring of Pan Enteric Mucosal Healing in Crohn's Disease Patients Treated With Vedolizumab
Brief Title: Pillcam Crohn's Capsule for Monitoring of Panenteric Mucosal Healing in Crohn's Disease Patients With Vedolizumab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Takeda (Industry); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-18-4710-UK-CTIL
Record Dates: First submitted 2019-03-17; First posted 2019-03-26 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: The patients are started on vedolizumab and are prospectively followed by capsule. There is no predefined intervention that stems from diagnostic observations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- all patients (Experimental): All enrolled patients- prospective observation (all patients are followed using videocapsule)
  Interventions: Other: prospective follow-up with videocapsule

INTERVENTIONS:
Other: prospective follow-up with videocapsule — prospective follow-up with videocapsule

SUMMARY:
The main aim of the study is to evaluate the lielihood of panenteric mucosal healing in Crohn's disease patients treated with vedolizumab The study will include patients with active Crohn's disease who are starting treatment with vedolizumab. The patients will undergo evaluation with panenteric capsule endoscopy, intestinal ultrasound and inflammatory biomarkers before treatment onset, at week 14 and week 52

DETAILED DESCRIPTION:
Mucosal healing has been widely accepted as the ultimate therapeutic goal in treatment of IBD patients and is associated with improved short and long-term outcomes in both ulcerative colitis and Crohn's disease (CD). However, the vast majority of the available clinical data pertains to colonic mucosal healing. In CD, the small bowel is involved in at least 75% of the patients, frequently in locations that are not accessible to ileocolonoscopy Active small bowel disease can be detected in at least 50% of CD patients in clinical remission[3]. Moreover, colonic and small bowel mucosal healing do not parallel each other, and it is quite common to detect inflammation in one segment while the other demonstrates endoscopically active disease.

Small bowel capsule endoscopy (SBCE) is the prime modality for evaluation of the entire small bowel[5]. It provides a safe and accurate way to screen and evaluate the entire small bowel, using a clinically validated endoscopic score such as the Lewis score (LS). Several studies evaluated the use of SBCE in monitoring mucosal healing in Crohn's disease, in both active and quiescent disease. The safety profile of SBCE in CD is excellent, especially after verification of small bowel patency using a patency capsule (PC).

To date, prospective data pertaining to the efficacy of biologics in induction of small bowel mucosal healing is very limited. The only prospective study to date was relatively small (36 patients) and demonstrated a significant improvement in mucosal inflammation and achievement of mucosal healing in patients that received Adalimumab and were evaluated with SBCE at week 0, 12 and 52 The rate of mucosal healing increased significantly from week 12 to 54.. No such data exists for other biologics. Recently, a combined pan-enteric capsule (PillCam Crohn's capsule) was developed by Medtronic. The capsule is based on an existing PillCam Colon 2 with a modified reading software. This capsule enables evaluation of mucosal inflammation and healing in the entire digestive tract in a single safe and non-invasive procedure. The new software of Rapid 9 includes a new method of describing the inflammatory burden on each of the 3 tertiles of the small bowel and two of the colon as well as the "old" Lewis score. In a feasibility 5 center prospective trial the capsule exited the colon while photographing in 83% of patients and reached the recto-sigma in 95%.

Intestinal ultrasound (IUS) is an accurate, safe and cheap modality for bedside evaluation of the small bowel. It was evaluated for both diagnosis and monitoring of intestinal inflammation in CD, and can be also utilized to assess the response to treatment. Recently, a quantitative score (Limberg index (LI)) for quantification of small bowel inflammation on IUS was validated.

The aim of our study is to assess the utility of the Pillcam Crohn's capsule in assessment of panenteric mucosal healing in CD patients treated with vedolizumab Study interventions

Visit 1 (before vedolizumab is started):

* Clinical activity
* Patients will perform patency capsule (PC) and give fecal sample for FC and microbiome.
* If PC is safely excreted within 30 hours and FC > 100 mg/kg, the patient will undergo SBC and will be enrolled if LS ≥ 220 or CDEIS>5.
* Blood will be drawn for measurement of CRP levels and complete blood count (CBC).
* IUS will be performed. Second visit and third visit(week 14 and 52): will include clinical evaluation, CBC, CRP, FCP, microbiome, SBC and IUS.

ELIGIBILITY:
Inclusion criteria:

* Crohn's disease
* planned to initiate VDZ treatment as recommended by the treating physician
* age- 18-70
* active small bowel inflammation on SBC (LS ≥ 220 or SES-CD>5 or active inflammation on the Pillcam Crohn's capsule score and FC>100 mg/kg)

Exclusion criteria:

* History of small bowel radiation
* History of previous capsule retention
* Previous treatment with vedolizumab

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Panenteric mucosal healing | 52 weeks
  Percentage of patients achieving pan enteric mucosal healing at week 52 post VDZ initiation as assessed by the Pillcam Crohn's capsule

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No